CLINICAL TRIAL: NCT06322901
Title: Examination Of The Effect Of Vertical Releasing Incision On Implant Procedures: A Randomized Controlled Split-Mouth Study
Brief Title: The Effect Of Vertical Releasing Incision On Implant Procedures
Acronym: Vertikal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Duygu Kilic, Dr, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: TDH-2018-7883
Record Dates: First submitted 2024-03-12; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Bone Loss; Flap Design
Keywords: flap design; vertical incision; OPG-RANKL; cortisol
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Surgical Flaps

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test side (Experimental): A mid-crestal incision was made on the test side with a no. 12 scalpel and a sulcular incision was made around the first natural tooth and a 5-mm vertical incision was made disto-obliquely to the distal crestal incision
  Interventions: Procedure: Flap
- control side (Active Comparator): Only a mid-crestal incision was made on the control side with a no. 12 scalpel and a sulcular incision was made around the first natural tooth
  Interventions: Procedure: Flap

INTERVENTIONS:
Procedure: Flap — Different flap designs for implant placement

SUMMARY:
This study evaluated the clinical and biochemical aspects of flap design in dental implant applications regarding implantation success and patient comfort. In this split-mouth randomized controlled clinical trial, a vertical releasing incision was made at the distal end of the crestal incision on the test side, and the control side received a crestal incision alone. Sixty-eight implants were placed in 17 patients. Peri-implant groove fluid was collected on postsurgical days 3, 7, 30, and 90; OPG and RANKL levels were assessed to determine bone formation and resorption around the implants. Cortisol levels were assessed in peri-implant groove fluid at postsurgical days 3, 7, and 14. Visual analog scale (VAS), and swelling measurements were taken postoperatively. Panoramic and periapical X-rays were obtained immediately post-surgery and at 3 months. No significant marginal bone loss difference was observed between the test and control sides at 3 months. The RANKL/OPG ratio, cortisol levels, VAS scores, and swelling scores were higher in the test vs. control sides. Overall, while the use of a vertical incision has advantages, such as increasing the visual field of the surgeon and improving the ease of the operation, this approach should be used only when necessary, given the disadvantages of increased bone resorption mediators in the peri-implant tissue and reduced postoperative patient comfort.

DETAILED DESCRIPTION:
Dental implantation is the most widely used method for treating edentulous patients. The most important factors affecting dental implant success are the patient's systemic condition, the material used, the physical properties of the implant, and the surgical protocol. Flap design is the first and most important stage of dental implant surgery. The most commonly used surgical technique for implant placement elevates the full-thickness mucoperiosteal flap. Flap design is critical in this procedure to reduce patient pain, limit stress-related cortisol level increases, and prevent peri-implant bone loss. An ideal flap reveals the entire surgical area, allowing the surgeon to work comfortably and place the implant in the desired position; thus, a vertical incision can be added to the flap. However, recent studies have demonstrated that a minimally invasive flap design reduces postoperative pain, bleeding, crestal bone loss, and surgical time. Several other studies concluded that flap designs with or without a vertical incision are equally successful.

Marginal bone resorption also influences long-term implantation success. Marginal bone resorption is aggravated by flap design and increases in cortisol secretion due to patient pain. High cortisol and β-endorphin concentrations can significantly increase MMP-1, MMP-2, MMP-7, MMP-11, and TIMP-1 levels in human gingival fibroblasts, explaining the increase in periodontal and peri-implant destruction associated with physiological stress. Several studies have offered acceptable explanations for the relationship between oral health (especially periodontal health) and psychological stres. The pathophysiological effects of periodontal disease are directly related to host resistance and affect the immune system. A positive relationship between salivary cortisol levels and stress levels has also been observed in individuals with severe periodontal disease. Marginal bone resorption around implants can be measured biochemically by examining substances in the peri-implant crevicular fluid, such as the markers osteoprotegerin (OPG) and receptor-activator NFkB ligand (RANKL). RANKL is a membrane-bound factor expressed on the outer surfaces of osteoblast cells and plays a central role in osteoclast cell formation and development. OPG binds to RANKL and prevents it from interacting with its receptor, NFkB, on osteoclasts and preosteoclasts, preventing bone loss. The OPG/RANKL ratio in the peri-implant groove fluid can indicate marginal bone resorption around dental implants; healthy implants demonstrate greater OPG/RANKL ratios than those with active marginal bone resorption. Thus, the effects of flap design on marginal bone loss (MBL) can be compared via the OPG/RANKL ratio.

Pain also causes systemic changes. The levels of cortisol, dehydroepiandrosterone, testosterone, and thyroid-stimulating hormone in bodily fluids can indicate a patient's pain level. Cortisol is controlled by adrenocorticotropic hormone (ACTH) released from the anterior pituitary gland. Most physical or neurological stressors strongly increase ACTH secretion, and dental stress increases bodily fluid hormone levels.

A literature review revealed insufficient studies examining the effects of a vertical incision on the peri-implant bone level. Existing studies only include clinical or radiological evaluations. This study aimed to evaluate the clinical effects of flap design and incision on dental implants by administering a visual analog scale (VAS) questionnaire, measuring swelling, recording the flap surgery duration, assessing the OPG/RANKL ratio and cortisol levels in the peri-implant groove fluid, and taking periapical X-ray images. Our study is unique and comprehensive since it addresses the clinical, biochemical, and radiological effects of a vertical incision on implants. In addition, although various studies have included cortisol measurements in the gingival crevicular fluid, few have measured cortisol in peri-implant groove fluid. Our findings suggest that flap designs with a vertical incision cause early marginal bone loss and additional stress on dental implant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral tooth deficiency in the lower jaw posterior region who received 2 dental implants on the right and left sides were recruited from the Erciyes University Faculty of Dentistry Department of Periodontology between December 2018 and January 2020

Exclusion Criteria:

* Patients were excluded if they had any systemic disease, demonstrated bone structure unsuitable for a 3.7 × 10 mm dental implant, were pregnant, had previously received radiotherapy or chemotherapy, had a tooth extracted from the implant area within 6 months, had active periodontal disease, required antibiotic prophylaxis, had inadequate keratinized gingiva, or demonstrated a tissue phenotype >2 mm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Bone loss | İnitial to 3rt mounth
  The degree of marginal bone loss (MBL) at the end of the 3rd month was determined and compared to the initial value. The following data were used to determine MBL: radiological marginal bone loss (RMBL), radiological implant length (RDİL), and real implant length (RİL).

OTHER OUTCOMES:
OPG/RANKL | days 3, 7, 14, 30, and 90
  OPG/RANKL in the peri-implant groove fluid were evaluated on postoperative days 3, 7, 14, 30, and 90
visual analog scale (VAS) | days 3, 7, and 14
  VAS (lowest = 0, highest 10) records were taken separately for the right and left sides of the lower jaw on postsurgical days 3, 7, and 14 to evaluate pain.
cortisol levels | days 3, 7, 14, 30, and 90
  cortisol levels in the peri-implant groove fluid were evaluated on postoperative days 3, 7, 14, 30, and 90

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Kılıç, Dr, Study Director — Erciyes University Faculty of Dentistry
Locations (1):
- Erciyes University Faculty of Dentistry, Melikgazi, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No